CLINICAL TRIAL: NCT04941781
Title: A Phase 1, Open-label Study of PIPE-307 to Determine Muscarinic Type I Receptor (M1AChR) Occupancy Parameters by [11C] PIPE-307 PET Imaging in Healthy Volunteers
Brief Title: PET Study to Determine the Relationship Between Plasma Concentrations and Muscarinic Type 1 Receptor (M1AChR) Occupancy of PIPE-307 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Contineum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTI-307-102
Record Dates: First submitted 2021-06-18; First posted 2021-06-28 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2021-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PIPE-307 (Experimental): Subjects will receive an oral dose of PIPE-307 and 3 intravenous injections of [11C] PIPE- 307.
  Interventions: Drug: PIPE-307

INTERVENTIONS:
Drug: PIPE-307 — Each dose cohort will receive a single oral dose of PIPE-307. Doses to be tested in subsequent cohorts will be determined by the analysis of the exposure from PK data and the PET scans with [11C] PIPE-307.
  Subjects will receive an intravenous dose of the radioligand [11C] PIPE-307 prior to PET imaging.

SUMMARY:
This is a Phase 1, single-center, open-label, adaptive-design PET study to investigate the occupancy of brain muscarinic Type 1 receptors (M1AChR) by PIPE-307 in healthy volunteers.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, open-label, adaptive-design study to investigate the occupancy of brain M1AChR after a single oral dose of PIPE-307 in healthy volunteers by positron emission tomography (PET) using the radioligand [11C] PIPE-307.

This study will have an adaptive design to adequately evaluate the relationship between PIPE-307 exposure and brain M1AChR occupancy.

ELIGIBILITY:
Key Criteria:

* Normotensive male or female volunteers between 25-65 years old
* Deemed healthy on the basis of a clinical history, physical examination, ECG, vital signs, and laboratory tests of blood and urine

Key Exclusion Criteria:

* Clinically relevant abnormal findings at the screening assessments
* Clinically relevant abnormal medical history or concurrent medical condition
* Acute or chronic illness
* Contraindications to MRI, CT, PET, or arterial cannulation procedures
* Significant exposure to research related radiation or other exposure (defined as ICRP category IIb or no more than 10 mSv)
* Positive tests for hepatitis B surface antigen (HBsAg) & Hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody
* Drug or alcohol abuse
* Smoke more than 10 cigarettes daily
* Loss of more than 400 mL blood
* Vital signs or ECGs outside the acceptable range

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
M1AChR receptor occupancy as determined by regional total volume of distribution (VT) of [11C] PIPE-307 at 24 hours | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom